CLINICAL TRIAL: NCT00158925
Title: The EASYTRAK EPI Clinical Investigation
Acronym: EASYTRAK EPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Clinicals0001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Bradycardia; Congestive Heart Failure
Keywords: Artificial Cardiac Pacing; Implanted Electrodes
MeSH Terms: conditions — Bradycardia; Heart Failure

ARMS (1):
- EASYTRAK EPI Lead (Experimental): Subjects in this arm will be implanted or attempted with the EASYTRAK EPI lead.
  Interventions: Device: EASYTRAK EPI lead

INTERVENTIONS:
Device: EASYTRAK EPI lead — EASYTRAK EPI lead

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of the EASYTRAK EPI lead.

DETAILED DESCRIPTION:
This is a prospective, single-armed, multi-center U.S., Australian, Canadian, and European clinical investigation, designed to demonstrate the safety and effectiveness of the EASYTRAK EPI lead in humans.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the EASYTRAK EPI indications
* Patients who are age 18 or above, or of legal age to give informed consent specific to state and national law
* Patients who are willing and capable of providing informed consent, undergoing a device implant, participating in all testing associated with this clinical investigation at an approved clinical investigational center and at the intervals defined by this protocol
* Patients who meet any one of the following three conditions:

  * Meet current indications for cardiac resynchronization therapy (CRT) and epicardial placement of a pace/sense lead on the left ventricle is preferred over an endocardial lead
  * Meet current indications for a cardiac pacing system and have documented evidence that an endocardial lead cannot be used
  * Meet current indications for a cardiac pacing system and a concurrent cardiac surgical procedure is taking place where no additional surgical procedures are required to provide access to the epicardial surface of the heart

Exclusion Criteria:

* Patients who meet the EASYTRAK EPI contraindications
* Patients who have had a myocardial infarct, unstable angina, or percutaneous coronary intervention during the preceding 30 days prior to enrollment
* Patients with a documented life expectancy of less than 6 months or expected to undergo heart transplant within the next 6 months
* Patients enrolled in any concurrent study, without Guidant written approval, that may confound the results of this study
* Women who are pregnant or plan to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Beckman, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Multiple Locations in the US, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EASYTRAK EPI Implant Group: This is a single arm study, all study subjects are to be implanted in 1 arm: the EASYTRAK EPI Implant Group.
Period: Overall Study
Arm/Group | EASYTRAK EPI Implant Group
Started | 96 (96 subjects were implanted or attempted with the study lead)
Completed | 84
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | EASYTRAK EPI Lead
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 74
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88
  Canada | 1
  Sweden | 7

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pacing Thresholds at 3 Months
Description: The expected mean pacing threshold is 1.9V at 0.5 ms pulse width.
Time Frame: 3 months
Population: Although 96 subjects were implanted/attempted, for 80 subjects still in follow up at the end of the 3M fu periodm the mean pacing threshold was obtained.
Measure: Mean (Standard Deviation); unit: V
Arm/Group | EASYTRAK EPI Implant Group
Number analyzed (Participants) | 80
V | 0.9 (0.5)

2. Primary Outcome: Chronic Pacing Impedances at 3 Months
Description: The expected mean impedance is 500 Ohms.
Time Frame: 3 months
Population: Although 96 subjects were implanted/attempted, for 80 subjects still in follow up at the end of the 3M fu period, the mean impedance was measured.
Measure: Mean (Standard Deviation); unit: Ohms
Arm/Group | EASYTRAK EPI Implant Group
Number analyzed (Participants) | 80
Ohms | 500 (137)

3. Primary Outcome: Chronic Sensing Amplitudes at 3 Months
Description: The expected mean is 10mV.
Time Frame: 3 months
Population: Although 96 subjects were implanted/attempted, for 67 subjects still in follow up at the end of the 3M fu period, chronic sensing amplitude was measured.
Measure: Mean (Standard Deviation); unit: mV
Arm/Group | EASYTRAK EPI Implant Group
Number analyzed (Participants) | 67
mV | 15.8 (7.2)

4. Primary Outcome: Lead-related Complication-free Rate at 3 Months
Description: The estimated target value for this endpoint is 80%.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: % of complication free-rate
Arm/Group | EASYTRAK EPI Implant Group
Number analyzed (Participants) | 96
% of complication free-rate | 97.9 [95.5 to 100]

5. Secondary Outcome: Lead Implant Time
Description: The estimated target value for average implant time is 30 minutes. Unit of measure will be the time period needed for the implant.
Time Frame: Implant
Population: Although 96 subjects were implanted/attempted, lead implant time was only collected for 69 subjects.
Measure: Mean (Standard Deviation); unit: h.min
Arm/Group | EASYTRAK EPI Implant Group
Number analyzed (Participants) | 69
h.min | 1.47 (1.05)

ADVERSE EVENTS:
Arm/Group | EASYTRAK EPI Implant Group
All-Cause Mortality (participants affected / at risk) | 15/96
Serious Adverse Events (participants affected / at risk) | 55/96
Other Adverse Events (participants affected / at risk) | 49/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EASYTRAK EPI Implant Group (N=96)
Unable to capture-LV (Cardiac disorders) | 2 (2)
Impedance>2000 Ohms LV lead (Cardiac disorders) | 1 (1)
Dislodgment-no reported signs-LV (Cardiac disorders) | 1 (1)
Dislodgment-multiple signs-LV (Cardiac disorders) | 1 (1)
Dislodgment-Unable to capture-LV (Cardiac disorders) | 3 (3)
Extracardiac stimulation-RV (Cardiac disorders) | 1 (1)
Infection (>30 days post implant) (Infections and infestations) | 2 (2)
Systemic infection (Infections and infestations) | 1 (1)
Post-up urinary retention (Renal and urinary disorders) | 2 (2)
Elevated blood glucose (Endocrine disorders) | 1 (1)
Hemorrhage-procedural related (Vascular disorders) | 1 (1)
Migration (Cardiac disorders) | 1 (1)
Thromboembolic events (Vascular disorders) | 3 (4)
Dehiscence of incision over PG (Surgical and medical procedures) | 1 (1)
Vasovagal symptoms (Vascular disorders) | 1 (1)
Post-surgical infection (<30 days post-implant) (Infections and infestations) | 3 (3)
Pneumothorax-procedure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma-pocket (Skin and subcutaneous tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Hypotension (Blood and lymphatic system disorders) | 4 (4)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Inadvertent VT/VF (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
General adverse reaction (General disorders) | 8 (12) — These adverse events were monitored/assessed without regard to the specific Adverse Event Term.
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (3)
Post-surgical wound-discomfort (Skin and subcutaneous tissue disorders) | 4 (4)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1)
Low cardiac output (Cardiac disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral vascular disease (Blood and lymphatic system disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 7 (10)
Gastrointestinal (Gastrointestinal disorders) | 6 (6)
Dyspnea (Cardiac disorders) | 3 (3)
Heart failure symptoms-unspecified (Cardiac disorders) | 4 (5)
Death (General disorders) | 2 (2)
Atelactasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Impedance > 2000 Ohms-RV lead (Cardiac disorders) | 1 (1)
Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Weight gain (Metabolism and nutrition disorders) | 2 (2)
Unable to capture- non RA lead related (Cardiac disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 4 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Peripheral edema (Blood and lymphatic system disorders) | 3 (3)
Cardiac arrest (Cardiac disorders) | 3 (3)
Urosepsis (Renal and urinary disorders) | 2 (2)
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1)
Chest pain-ischemic (Cardiac disorders) | 1 (1)
Physical trauma (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Cardiac disorders) | 1 (1)
Abnormal lab values (Blood and lymphatic system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Multi-system failure (Cardiac disorders) | 3 (3)
Endocrine (Endocrine disorders) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (3)
Tooth extraction (Surgical and medical procedures) | 1 (2)
Aortic stenosis (Cardiac disorders) | 1 (1)
Thrombus (Blood and lymphatic system disorders) | 1 (1)
Distal thromboemboli (Blood and lymphatic system disorders) | 1 (1)
Pulmonary symtpoms (Respiratory, thoracic and mediastinal disorders) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EASYTRAK EPI Implant Group (N=96)
General adverse event (General disorders) | 11 (14) — Adverse events were monitored/assessed without regard to the specific Adverse Event Term.
Atrial fibrillation (Cardiac disorders) | 10 (12)
Extracardiac stimulation-LV lead (Cardiac disorders) | 6 (8)
Hypotension (Blood and lymphatic system disorders) | 5 (5)
Inappropriate tachy therapy (Cardiac disorders) | 5 (5)
Post-surgical wound discomfort (Skin and subcutaneous tissue disorders) | 6 (8)
Pulmonary adverse events (Respiratory, thoracic and mediastinal disorders) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other